CLINICAL TRIAL: NCT01669434
Title: Chronic Angiotensin Converting Enzyme Inhibitors in Intermediate Risk Surgery: A Randomized, Single-Blinded Study
Brief Title: Chronic Angiotensin Converting Enzyme Inhibitors in Intermediate Risk Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0369-12-FB
Record Dates: First submitted 2012-08-14; First posted 2012-08-21 (Estimated); Results first posted 2017-12-11 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Hypotension on Induction
Keywords: Perioperative Period
MeSH Terms: interventions — Quinapril; Perindopril; Ramipril; benazepril; Captopril; Enalapril; Enalaprilat; Fosinopril; Lisinopril; trandolapril; moexipril

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ACEI continuation (Experimental): Patients in this arm will be randomized to continue their chronic angiotensin converting enzyme inhibitor without interruption preoperatively
  Interventions: Drug: ACEI continuation
- ACEI omission (Experimental): Patients randomized to this arm will be told to omit their final preoperative chronic angiotensin converting enzyme inhibitor dose.
  Interventions: Drug: ACEI omission

INTERVENTIONS:
Drug: ACEI continuation — These chronic medications will be taken without interruption preoperatively.
  Other Names: quinapril; Accupril; perindopril; Aceon; ramipril; Altace; benazepril; Lotensin; captopril; Capoten; enalapril; Vasotec; fosinopril; Monopril; lisinopril; Prinivil; Zestril; trandolapril; Mavik; moexipril; Univasc
  Arms: ACEI continuation
Drug: ACEI omission — Although taken chronically by patients in this intervention, the final preoperative dose of these medications will be omitted, whether it was scheduled for the morning of surgery or the day prior.
  Other Names: quinapril; Accupril; perindopril; Aceon; ramipril; Altace; benazepril; Lotensin; captopril; Capoten; enalapril; Vasotec; fosinopril; Monopril; lisinopril; Prinivil; Zestril; trandolapril; Mavik; moexipril; Univasc
  Arms: ACEI omission

SUMMARY:
Primary research hypothesis: Patients who continue their chronic ACEI therapy up to and including the morning of a non-cardiac, non-vascular surgery will experience more intraoperative hypotension than those who transiently hold their chronic ACEI preoperatively.

Secondary research hypothesis #1: Patients who continue their chronic ACEI up to and including the morning of a non-cardiac, non-vascular surgery will experience better postoperative control of hypertension than those who transiently hold their chronic ACEI preoperatively.

Secondary research hypothesis #2: Patients who continue their chronic ACEI up to and including the morning of a non-cardiac, non-vascular surgery will experience less acute renal failure than those who transiently hold their chronic ACEI preoperatively.

Secondary research hypothesis #3: In the subgroup of patients with a preoperative systolic blood pressure less than 110 mmHg, those who continue their chronic ACEI therapy up to and including the morning of a non-cardiac, non-vascular surgery will experience more intraoperative hypotension than those who transiently hold their chronic ACEI preoperatively.

Secondary research hypothesis #4: In the subgroup of patients above the age of 64, those who continue their chronic ACEI therapy up to and including the morning of a non-cardiac, non-vascular surgery will experience more intraoperative hypotension than those who transiently hold their chronic ACEI preoperatively.

DETAILED DESCRIPTION:
The purpose of this study is to determine if transient discontinuation of angiotensin converting enzyme inhibitors (ACEIs) is necessary prior to non-cardiac, non-vascular surgery. ACEIs have been associated with intraoperative hypotension during vascular and cardiac surgeries. Patients presenting to the University of Nebraska Medical Center Pre-Anesthesia Screening (PAS) Clinic who are on chronic ACEI therapy will be eligible for enrollment. Subjects will be randomized to either omit or continue their ACEI preoperatively. The outcome of interest is intraoperative hypotension defined as a systolic blood pressure less than 80 mmHg. Blood pressure will be followed not only throughout surgery, but also during recovery and the remainder of hospitalization. Renal function will be assessed with creatinine measurements in the PAS clinic and on the first postoperative day. No follow-up is planned beyond discharge from the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Referred to the University of Nebraska Medical Center Pre-Anesthesia Screening Clinic for preoperative evaluation.
* Above referral must be in anticipation of a non-cardiac, non-vascular surgery.
* Must have been on ACE-Inhibitor therapy for at least six weeks.

Exclusion Criteria:

* Hypotension (systolic blood pressure < 90 or diastolic blood pressure <60) at the time of preoperative evaluation
* Uncontrolled Hypertension (systolic blood pressure > 150 or diastolic blood pressure > 95) at the time of preoperative evaluation
* Surgery during which vasopressor use is anticipated (carotid endarterectomy, major abdominal operations, orthopedic oncology)
* Surgery for pathology related to vasoactive substances (carcinoid, pheochromocytoma)
* Left Ventricular ejection fraction less than 40%
* Clinical evidence of decompensated heart failure at the time of preoperative evaluation
* End-stage renal disease
* Organ transplant surgeries

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 291 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2016-11-01 (Actual); Study Completion 2016-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason F Shiffermiller, MD, MPH, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McConachie I, Healy TE. ACE inhibitors and anaesthesia. Postgrad Med J. 1989 May;65(763):273-4. doi: 10.1136/pgmj.65.763.273. No abstract available. PMID 2692007
- [Background] Coriat P, Richer C, Douraki T, Gomez C, Hendricks K, Giudicelli JF, Viars P. Influence of chronic angiotensin-converting enzyme inhibition on anesthetic induction. Anesthesiology. 1994 Aug;81(2):299-307. doi: 10.1097/00000542-199408000-00006. PMID 8053578
- [Background] Comfere T, Sprung J, Kumar MM, Draper M, Wilson DP, Williams BA, Danielson DR, Liedl L, Warner DO. Angiotensin system inhibitors in a general surgical population. Anesth Analg. 2005 Mar;100(3):636-644. doi: 10.1213/01.ANE.0000146521.68059.A1. PMID 15728043
- [Background] Pigott DW, Nagle C, Allman K, Westaby S, Evans RD. Effect of omitting regular ACE inhibitor medication before cardiac surgery on haemodynamic variables and vasoactive drug requirements. Br J Anaesth. 1999 Nov;83(5):715-20. doi: 10.1093/bja/83.5.715. PMID 10690132
- [Background] Steiner CA, Karaca Z, Moore BJ, Imshaug MC, Pickens G. Surgeries in Hospital-Based Ambulatory Surgery and Hospital Inpatient Settings, 2014. 2017 May [updated 2020 Jul 20]. In: Healthcare Cost and Utilization Project (HCUP) Statistical Briefs [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2006 Feb-. Statistical Brief #223. Available from http://www.ncbi.nlm.nih.gov/books/NBK442035/ PMID 28722845
- [Background] Rate of all-listed procedures for discharges from short-stay hospitals, by procedure category and age: United States, 2010. 2010.
- [Background] Turan A, You J, Shiba A, Kurz A, Saager L, Sessler DI. Angiotensin converting enzyme inhibitors are not associated with respiratory complications or mortality after noncardiac surgery. Anesth Analg. 2012 Mar;114(3):552-60. doi: 10.1213/ANE.0b013e318241f6af. Epub 2012 Jan 17. PMID 22253266
- [Background] Mascha EJ, Yang D, Weiss S, Sessler DI. Intraoperative Mean Arterial Pressure Variability and 30-day Mortality in Patients Having Noncardiac Surgery. Anesthesiology. 2015 Jul;123(1):79-91. doi: 10.1097/ALN.0000000000000686. PMID 25929547
- [Background] Walsh M, Devereaux PJ, Garg AX, Kurz A, Turan A, Rodseth RN, Cywinski J, Thabane L, Sessler DI. Relationship between intraoperative mean arterial pressure and clinical outcomes after noncardiac surgery: toward an empirical definition of hypotension. Anesthesiology. 2013 Sep;119(3):507-15. doi: 10.1097/ALN.0b013e3182a10e26. PMID 23835589
- [Background] Bertrand M, Godet G, Meersschaert K, Brun L, Salcedo E, Coriat P. Should the angiotensin II antagonists be discontinued before surgery? Anesth Analg. 2001 Jan;92(1):26-30. doi: 10.1097/00000539-200101000-00006. PMID 11133595
- [Background] Roshanov PS, Rochwerg B, Patel A, Salehian O, Duceppe E, Belley-Cote EP, Guyatt GH, Sessler DI, Le Manach Y, Borges FK, Tandon V, Worster A, Thompson A, Koshy M, Devereaux B, Spencer FA, Sanders RD, Sloan EN, Morley EE, Paul J, Raymer KE, Punthakee Z, Devereaux PJ. Withholding versus Continuing Angiotensin-converting Enzyme Inhibitors or Angiotensin II Receptor Blockers before Noncardiac Surgery: An Analysis of the Vascular events In noncardiac Surgery patIents cOhort evaluatioN Prospective Cohort. Anesthesiology. 2017 Jan;126(1):16-27. doi: 10.1097/ALN.0000000000001404. PMID 27775997
- [Background] Fleisher LA, Fleischmann KE, Auerbach AD, Barnason SA, Beckman JA, Bozkurt B, Davila-Roman VG, Gerhard-Herman MD, Holly TA, Kane GC, Marine JE, Nelson MT, Spencer CC, Thompson A, Ting HH, Uretsky BF, Wijeysundera DN; American College of Cardiology; American Heart Association. 2014 ACC/AHA guideline on perioperative cardiovascular evaluation and management of patients undergoing noncardiac surgery: a report of the American College of Cardiology/American Heart Association Task Force on practice guidelines. J Am Coll Cardiol. 2014 Dec 9;64(22):e77-137. doi: 10.1016/j.jacc.2014.07.944. Epub 2014 Aug 1. No abstract available. PMID 25091544
- [Background] Kristensen SD, Knuuti J, Saraste A, Anker S, Botker HE, Hert SD, Ford I, Gonzalez-Juanatey JR, Gorenek B, Heyndrickx GR, Hoeft A, Huber K, Iung B, Kjeldsen KP, Longrois D, Luscher TF, Pierard L, Pocock S, Price S, Roffi M, Sirnes PA, Sousa-Uva M, Voudris V, Funck-Brentano C; Authors/Task Force Members. 2014 ESC/ESA Guidelines on non-cardiac surgery: cardiovascular assessment and management: The Joint Task Force on non-cardiac surgery: cardiovascular assessment and management of the European Society of Cardiology (ESC) and the European Society of Anaesthesiology (ESA). Eur Heart J. 2014 Sep 14;35(35):2383-431. doi: 10.1093/eurheartj/ehu282. Epub 2014 Aug 1. No abstract available. PMID 25086026
- [Background] Mehta RL, Kellum JA, Shah SV, Molitoris BA, Ronco C, Warnock DG, Levin A; Acute Kidney Injury Network. Acute Kidney Injury Network: report of an initiative to improve outcomes in acute kidney injury. Crit Care. 2007;11(2):R31. doi: 10.1186/cc5713. PMID 17331245
- [Background] Monk TG, Bronsert MR, Henderson WG, Mangione MP, Sum-Ping ST, Bentt DR, Nguyen JD, Richman JS, Meguid RA, Hammermeister KE. Association between Intraoperative Hypotension and Hypertension and 30-day Postoperative Mortality in Noncardiac Surgery. Anesthesiology. 2015 Aug;123(2):307-19. doi: 10.1097/ALN.0000000000000756. PMID 26083768
- [Background] Kheterpal S, Khodaparast O, Shanks A, O'Reilly M, Tremper KK. Chronic angiotensin-converting enzyme inhibitor or angiotensin receptor blocker therapy combined with diuretic therapy is associated with increased episodes of hypotension in noncardiac surgery. J Cardiothorac Vasc Anesth. 2008 Apr;22(2):180-6. doi: 10.1053/j.jvca.2007.12.020. PMID 18375317
- [Background] Twersky RS, Goel V, Narayan P, Weedon J. The risk of hypertension after preoperative discontinuation of angiotensin-converting enzyme inhibitors or angiotensin receptor antagonists in ambulatory and same-day admission patients. Anesth Analg. 2014 May;118(5):938-44. doi: 10.1213/ANE.0000000000000076. PMID 24681657
- [Background] Tan TW, Eslami MH, Kalish JA, Eberhardt RT, Doros G, Goodney PP, Cronenwett JL, Farber A; Vascular Study Group of New England. The need for treatment of hemodynamic instability following carotid endarterectomy is associated with increased perioperative and 1-year morbidity and mortality. J Vasc Surg. 2014 Jan;59(1):16-24.e1-2. doi: 10.1016/j.jvs.2013.07.025. Epub 2013 Aug 30. PMID 23994095
- [Background] Lee SM, Takemoto S, Wallace AW. Association between Withholding Angiotensin Receptor Blockers in the Early Postoperative Period and 30-day Mortality: A Cohort Study of the Veterans Affairs Healthcare System. Anesthesiology. 2015 Aug;123(2):288-306. doi: 10.1097/ALN.0000000000000739. PMID 26200181
- [Background] Drenger B, Fontes ML, Miao Y, Mathew JP, Gozal Y, Aronson S, Dietzel C, Mangano DT; Investigators of the Ischemia Research and Education Foundation; Multicenter Study of Perioperative Ischemia Research Group. Patterns of use of perioperative angiotensin-converting enzyme inhibitors in coronary artery bypass graft surgery with cardiopulmonary bypass: effects on in-hospital morbidity and mortality. Circulation. 2012 Jul 17;126(3):261-9. doi: 10.1161/CIRCULATIONAHA.111.059527. Epub 2012 Jun 19. PMID 22715473
- [Derived] Shiffermiller JF, Monson BJ, Vokoun CW, Beachy MW, Smith MP, Sullivan JN, Vasey AJ, Guda P, Lyden ER, Ellis SJ, Pang H, Thompson RE. Prospective Randomized Evaluation of Preoperative Angiotensin-Converting Enzyme Inhibition (PREOP-ACEI). J Hosp Med. 2018 Sep;13(10):661-667. doi: 10.12788/jhm.3036. Epub 2018 Jul 25. PMID 30261084

RESULTS

PARTICIPANT FLOW:
Groups:
- ACEI Omission: Patients randomized to this arm will be told to hold their final preoperative angiotensin converting enzyme inhibitor dose.
  ACEI omission: These medications, although taken chronically by patients in this intervention, will not be given on the morning of surgery or day before surgery, whenever the last preoperative dose would normally occur.
- ACEI Continuation: Patients in this arm will be randomized to take their final preoperative angiotensin converting enzyme inhibitor dose.
  ACEI continuation: These chronic medications will be given without interruption preoperatively.
Period: Overall Study
Arm/Group | ACEI Omission | ACEI Continuation
Started | 146 | 145
Completed | 137 | 138
Not Completed | 9 | 7

BASELINE CHARACTERISTICS:
Groups:
- ACEI Omission: Patients randomized to this arm will be told to hold their final preoperative angiotensin converting enzyme inhibitor dose.
  ACEI omission: These medications, although taken chronically by patients in this intervention, will not be given on the morning of surgery or evening before surgery, whenever the last preoperative dose would normally occur.
- Total: Total of all reporting groups
Arm/Group | ACEI Omission | ACEI Continuation | Total
Number analyzed (Participants) | 137 | 138 | 275
Age, Continuous [Mean (Full Range); unit: years] | 64 [26 to 91] | 63.7 [31 to 86] | 63.9 [26 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 70 | 142
  Male | 65 | 68 | 133
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 115 | 125 | 240
  Black | 15 | 11 | 26
  Hispanic | 2 | 0 | 2
  Am Indian/Alaska | 2 | 1 | 3
  Other/Unknown | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 137 | 138 | 275
smoking status [Count of Participants; unit: Participants]
  Never | 63 | 54 | 117
  Former | 60 | 59 | 119
  Current | 14 | 25 | 39
American Society of Anesthesiologists classification [Mean (Full Range); unit: units on a scale] — Scale range 1-6 I A normal healthy patient Healthy, non-smoking, no or minimal alcohol use 2 A patient with mild systemic disease 3 A patient with severe systemic disease 4 A patient with severe systemic disease that is a constant threat to life 5 A moribund patient who is not expected to survive without the operation 6 A declared brain-dead patient whose organs are being removed for donor purposes
  units on a scale | 2.8 [1 to 4] | 2.8 [2 to 4] | 2.8 [1 to 4]
preoperative NSAID use [Count of Participants; unit: Participants] | 53 | 71 | 124
preoperative systolic BP [Mean (Full Range); unit: mmHg] | 136.6 [99 to 187] | 136.3 [102 to 184] | 136.5 [99 to 187]
hypertension history [Count of Participants; unit: Participants] | 116 | 112 | 228
congestive heart failure history [Count of Participants; unit: Participants] | 7 | 9 | 16
Additional antihypertensive [Count of Participants; unit: Participants] — Use of at least one additional antihypertensive medication in addition to an angiotensin converting enzyme inhibitor at the time of enrollment.
  Participants | 92 | 95 | 187

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Interoperative Hypotension
Description: Number of Participants with Interoperative Hypotension (systolic blood pressure under 80 mmHg)
Time Frame: During anesthesia, an expected average of 3 hours.
Measure: Count of Participants; unit: Participants
Arm/Group | ACEI Omission | ACEI Continuation
Number analyzed (Participants) | 137 | 138
Participants | 76 | 95
Statistical Analysis 1: Comparison: ACEI Omission vs ACEI Continuation; Test type: Superiority; p = 0.03, Fisher Exact; Risk Ratio (RR) = 0.81, 95% CI 2-sided [0.67 to 0.97]

2. Secondary Outcome: Acute Renal Failure
Description: Creatinine increase of more than 0.3 mg/dl or more than 50% from preoperative level
Time Frame: Arrival in post-anesthesia care unit (PACU) to hospital discharge, an expected average of 4 days.
Population: Missing outcome data for 37 patients, 18 in the ACEI omission arm and 19 in the ACEI continuation arm
Measure: Count of Participants; unit: Participants
Arm/Group | ACEI Omission | ACEI Continuation
Number analyzed (Participants) | 119 | 119
Participants | 6 | 10
Statistical Analysis 1: Comparison: ACEI Omission vs ACEI Continuation; Test type: Superiority; p = 0.44, Fisher Exact; Risk Ratio (RR) = 0.60, 95% CI 2-sided [0.23 to 1.60]

3. Secondary Outcome: Low Blood Pressure Subgroup
Description: Only patients with systolic blood pressure less than 110 at preoperative evaluation will be included in this analysis. The outcome is the same as the primary outcome: Intraoperative Systolic Blood Pressure under 80 mmHg.
Time Frame: During anesthesia, an expected average of 3 hours.
Measure: Count of Participants; unit: Participants
Arm/Group | ACEI Omission | ACEI Continuation
Number analyzed (Participants) | 5 | 3
Participants | 4 | 2
Statistical Analysis 1: Comparison: ACEI Omission vs ACEI Continuation; Test type: Superiority; p = 1.0, Fisher Exact; Risk Ratio (RR) = 1.20, 95% CI 2-sided [0.48 to 2.99]

4. Secondary Outcome: Older Age Subgroup
Description: Only patients above the age of 64 will be included in this analysis. The outcome is the same as the primary outcome: Intraoperative Systolic Blood Pressure under 80 mmHg
Time Frame: During anesthesia, an expected average of 3 hours.
Measure: Count of Participants; unit: Participants
Arm/Group | ACEI Omission | ACEI Continuation
Number analyzed (Participants) | 70 | 72
Participants | 48 | 49
Statistical Analysis 1: Comparison: ACEI Omission vs ACEI Continuation; Test type: Superiority; p = 1.0, Fisher Exact; Risk Ratio (RR) = 1.01, 95% CI 2-sided [0.81 to 1.26]

5. Secondary Outcome: Postoperative Hypertension
Description: Any systolic blood pressure greater than 180 mmHg.
Time Frame: Arrival in PACU to hospital discharge, an expected average of 4 days.
Measure: Count of Participants; unit: Participants
Arm/Group | ACEI Omission | ACEI Continuation
Number analyzed (Participants) | 137 | 138
Participants | 33 | 17
Statistical Analysis 1: Comparison: ACEI Omission vs ACEI Continuation; Test type: Superiority; p = 0.01, Fisher Exact; Risk Ratio (RR) = 1.95, 95% CI 2-sided [1.14 to 3.34]

6. Secondary Outcome: Postoperative Hypotension
Description: Any systolic blood pressure less than 90 mmHg
Time Frame: Arrival in PACU to hospital discharge, an expected average of 4 days.
Measure: Count of Participants; unit: Participants
Arm/Group | ACEI Omission | ACEI Continuation
Number analyzed (Participants) | 137 | 138
Participants | 15 | 31
Statistical Analysis 1: Comparison: ACEI Omission vs ACEI Continuation; Test type: Superiority; p = 0.02, Fisher Exact; Risk Ratio (RR) = 0.49, 95% CI 2-sided [0.28 to 0.86]

ADVERSE EVENTS:
Time Frame: Hospitalization, expected duration 4 days
Arm/Group | ACEI Omission | ACEI Continuation
All-Cause Mortality (participants affected / at risk) | 0/137 | 0/138
Serious Adverse Events (participants affected / at risk) | 4/137 | 1/138
Other Adverse Events (participants affected / at risk) | 0/137 | 0/138
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ACEI Omission (N=137) | ACEI Continuation (N=138)
MACE (Cardiac disorders) | 4 (4) | 1 (1) — Major Adverse Cardiac Event. A composite of acute coronary syndrome, acute heart failure, or new-onset arrhythmia

LIMITATIONS AND CAVEATS:
Management decisions were made by the treatment which was not blinded to allocation; Intraoperative hypotension is an intermediate measure but one that has known associations with adverse outcomes, including mortality.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No